CLINICAL TRIAL: NCT03920046
Title: Effects of Passive Smoking on Children During Gastrointestinal Endoscopy
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sibel Seçkin Pehlivan, Teaching Assistant, TC Erciyes University
Other Study IDs: 2018/641
Record Dates: First submitted 2019-04-08; First posted 2019-04-18 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Gastro-Intestinal Disorders
Keywords: esophagogastroduodenoscopy; laryngospasm; passive smoking; sedation
MeSH Terms: conditions — Laryngismus | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Effects of passive smoking on children: The prevalence of laryngospasm in sedation applied to endoscopic intervention whose parents smoking.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Control Group — The prevalence of laryngospasm in sedation applied to endoscopic intervention whose parents no smoking.

SUMMARY:
To evaluate the effect of passive smoking in children during Gastrointestinal Endoscopy.

DETAILED DESCRIPTION:
When the patients and their parents are arrived in the endoscopy unıt about 1 h before the procedure, the anesthetist is obtained a medical history and carried out a physical examination and clinical assesment. Then the parents smoking habits are documented about to detect the magnitude of passive smoking. Endoscopist and anesthesiologist are blinded to the patients passive smoking history. Then the sedation is applied and esophagogastroduodenoscopy procedures performed. Side effects (e.g laryngospasm, coughing) during the study are recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA ( American Society of Anesthesiologists) I- ASA II patients
* Aged 1- 18 Year old patients

Exclusion Criteria:

* Smoker patients

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Esophagogastroduodenoscopy patients are included in the study
Sampling Method: Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
laryngospasm ratio | an average of 2 hours
  The prevalence of laryngospasm in sedation applied to endoscopic intervention whose parents smoking.

SECONDARY OUTCOMES:
hypoxia ratio (oxygen saturation < % 90) | an average of 2 hours
  The prevalence of hypoxia (oxygen saturation < % 90) in sedation applied to endoscopic intervention whose parents smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- Sibel Seçkin Pehlivan, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De- identified individual participant data for all primary and secondary outcome measures will be available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 36 months of study completion.
Access Criteria: Data accept requests will be reviewed by an external independent Review Panel.Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Chung HK, Lightdale JR. Sedation and Monitoring in the Pediatric Patient during Gastrointestinal Endoscopy. Gastrointest Endosc Clin N Am. 2016 Jul;26(3):507-25. doi: 10.1016/j.giec.2016.02.004. PMID 27372774
- [Result] Rodrigo C. The effects of cigarette smoking on anesthesia. Anesth Prog. 2000 Winter;47(4):143-50. PMID 11432181
- [Result] Tosun Z, Aksu R, Guler G, Esmaoglu A, Akin A, Aslan D, Boyaci A. Propofol-ketamine vs propofol-fentanyl for sedation during pediatric upper gastrointestinal endoscopy. Paediatr Anaesth. 2007 Oct;17(10):983-8. doi: 10.1111/j.1460-9592.2007.02206.x. PMID 17767636
- [Derived] Pehlivan SS, Gergin OO, Bayram A, Altay D, Arslan D, Bicer C, Aksu R. The effect of passive smoking on the laryngospasm rate in children sedated during the esophagogastroduodenoscopy. Saudi Med J. 2022 Mar;43(3):275-282. doi: 10.15537/smj.2022.43.3.20210784. PMID 35256495